CLINICAL TRIAL: NCT00409006
Title: A Phase 2 Trial of Pemetrexed and Cisplatin Followed Sequentially by Gefitinib Versus Pemetrexed and Cisplatin in Asian "Never Smoker" Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Chemotherapy for Patients With Non-Small Cell Lung Cancer Who Are Non-Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10918; H3E-AA-S110 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Cisplatin/Gefitinib (Experimental): Pemetrexed 500 milligrams per meters squared (mg/m2) plus cisplatin 75 mg/m2 administered by intravenous (IV) infusion once every 3 weeks for 4 cycles without progression followed by gefitinib 250 mg administered orally, once daily, until disease progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Gefitinib
- Pemetrexed/Cisplatin (Experimental): Pemetrexed 500 milligrams per meters squared (mg/m2) plus cisplatin 75 mg/m2 administered by intravenous (IV) infusion once every 3 weeks for 4 cycles without progression followed by pemetrexed 500 mg/m2 administered by IV infusion (with optional cisplatin 75 mg/m2 for up to 2 additional cycles) until disease progression or unacceptable toxicity.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 milligrams per meter squared (mg/m2), administered by intravenous (IV) infusion every 21 days for 4 cycles (1-4) or 500 mg/m2, IV, every 21 days until disease progression or unacceptable toxicity.
  Other Names: LY231514; Alimta
Drug: Cisplatin — 75 mg/m2, IV, every 21 days for 4 cycles (1-4) or 75 mg/m2, IV, every 21 days for 4 cycles with optional continuation for 2 additional cycles until disease progression or unacceptable toxicity
Drug: Gefitinib — 250 mg, administered orally once daily beginning at Cycle 5 until disease progression or unacceptable toxicity
  Arms: Pemetrexed/Cisplatin/Gefitinib

SUMMARY:
The purpose of this study is to compare the efficacy and safety of chemotherapy followed sequentially by gefitinib versus chemotherapy alone in the first line treatment of non-small cell lung cancer (NSCLC). This study will be conducted in Asian patients who are classified as 'never smoker' since it is suggested that these patients are more likely to respond favorably to treatment with gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis non-small cell lung cancer (NSCLC) (Stage IIIB or IV)
* Have not received any prior chemotherapy, molecular therapy, immunotherapy, biological therapy, or radiotherapy. Exception: palliative radiotherapy that is completed at least 4 weeks prior to study enrolment.
* Have 'never smoked' (defined as having smoked <100 cigarettes during his/her lifetime)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1

Exclusion Criteria:

* Concurrent administration of any other tumor therapy
* Other co-existing malignancies
* Pregnancy or breast feeding
* Serious concomitant disorders
* Inability or unwillingness to take folic acid or vitamin B12 supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fujian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Qingdao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

REFERENCES:
- [Derived] Ahn MJ, Yang JC, Liang J, Kang JH, Xiu Q, Chen YM, Blair JM, Peng G, Linn C, Orlando M. Randomized phase II trial of first-line treatment with pemetrexed-cisplatin, followed sequentially by gefitinib or pemetrexed, in East Asian, never-smoker patients with advanced non-small cell lung cancer. Lung Cancer. 2012 Aug;77(2):346-52. doi: 10.1016/j.lungcan.2012.03.011. Epub 2012 Apr 23. PMID 22534669
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 86 participants entered study. 13 participants were screen failures. 73 participants (40 pemetrexed/cisplatin/gefitinib and 33 pemetrexed/cisplatin) were assigned to treatment. 3 participants did not receive study drug. These 16 participants (13 screen failures and 3 that did not receive drug) were not included in the analyses.
Period: Overall Study
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Started | 39 | 31
Completed | 19 | 19
Not Completed | 20 | 12
Not completed — Death | 15 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin | Total
Number analyzed (Participants) | 39 | 31 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 55.6 (8.45) | 55.7 (12.43) | 55.7 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  East Asian | 39 | 31 | 70
Region of Enrollment [Number; unit: participants]
  Taiwan | 10 | 11 | 21
  China | 16 | 14 | 30
  Korea, Republic of | 13 | 6 | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Units on a scale] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death). 0 - Fully Active. 1 - Ambulatory, Restricted Strenuous Activity. 2 - Ambulatory, No Work Activities. 3 - Partially Confined to Bed, Limited Self Care. 4 - Completely Disabled.
  Units on a scale
    0 | 15 | 9 | 24
    1 | 24 | 22 | 46
History of Smoking [Number; unit: Participants]
  Yes | 0 | 2 | 2
  No | 39 | 29 | 68
Basis of Diagnosis [Number; unit: Participants]
  Histopathological | 30 | 22 | 52
  Cytological | 9 | 9 | 18
Pathological Diagnosis [Number; unit: Participants]
  Mixed Cell Carcinoma, Lung | 1 | 1 | 2
  Adenocarcinoma | 30 | 24 | 54
  Carcinoma, Squamous Cell | 7 | 4 | 11
  Non-Small Cell Lung Carcinoma | 1 | 2 | 3
Disease Stage [Number; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage 0 - the cancer has not spread beyond the inner lining of the lung. Stage I - the cancer is small and hasn't spread to the lymph nodes. Stage II - the cancer has spread to some lymph nodes near the original tumor. Stage III - the cancer has spread to nearby tissue or spread to far away lymph nodes. Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  Participants
    Stage IIIB | 6 | 4 | 10
    Stage IV | 33 | 27 | 60

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from randomization to the first observation of disease progression, or death due to any cause.
Time Frame: Baseline to first observation of disease progression or death, 12 weeks up to 31 months
Population: Randomized and treated (RT) population includes all randomized patients. Patients are analyzed according to the treatment they actually received (intent-to-treat [ITT] analysis). Patients were censored from this analysis (8 pemetrexed/cisplatin/gefitinib and 11 pemetrexed/cisplatin).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 31
Months | 9.95 [5.85 to 16.49] | 6.83 [5.78 to 7.98]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin/Gefitinib vs Pemetrexed/Cisplatin; Test type: Superiority or Other; p = 0.0618, Log Rank

2. Secondary Outcome: Number of Participants With Tumor Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes not meeting above criteria. Responder is a participant exhibiting a best overall study response of CR or PR.
Time Frame: Baseline to measured response or death, 12 weeks up to 31 months
Population: Qualified for Response population includes all treated patients with measurable disease prior first dose of study therapy.
Measure: Number; unit: Participants
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 31
Participants | 18 [30.1 to 62.8] | 11 [19.2 to 54.6]
Statistical Analysis 1: Comparison: Pemetrexed/Cisplatin/Gefitinib vs Pemetrexed/Cisplatin; Test type: Superiority or Other; p = 0.369, Regression, Logistic; Used the Wald Chi-squared statistic from a logistic regression analysis

3. Secondary Outcome: Duration of Response for Responders
Description: The duration of a complete response (CR; the disappearance of all target lesions) or partial response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause. A responder is a patient exhibiting a best overall study response of CR or PR.
Time Frame: Time of response to progressive disease or death, 12 weeks up to 31 months
Population: Qualified for Response population includes all treated patients with measurable disease prior first dose of study therapy. Patients were censored for this analysis (2 pemetrexed/cisplatin/gefitinib and 2 pemetrexed/cisplatin).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Number analyzed (Participants) | 18 | 11
Months | 12.29 [8.51 to 15.31] | 4.14 [2.76 to 7.62]

4. Post Hoc Outcome: Percentage of Participants Who Died During the Study
Description: This outcome measure takes the place of the outcome measure for Overall Survival, which could not be reported since the median value could not be calculated.
Time Frame: Baseline up to 31 months
Population: Randomized and treated population includes all randomized patients. Patients are analyzed according to the treatment they actually received (ITT population). 25 participants from each treatment group were censored.
Measure: Number; unit: Percentage of Participants
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Number analyzed (Participants) | 39 | 31
Percentage of Participants | 35.9 | 19.4

5. Secondary Outcome: Overall Survival
Description: Overall survival is the duration from enrollment to death. For patients who are alive, overall survival is censored at the last contact. Median overall survival could not be estimated as most participants were living at the end of the study. 25 participants from each treatment group were censored. In place of this outcome measure, the percentage of participants who died during the study are provided in the Post-Hoc Analysis Outcome Measure: Percentage of Participants Who Died During the Study.
Time Frame: Baseline to date of death from any cause, 12 weeks up to 31 months
Population: Randomized and treated population includes all randomized patients. Patients are analyzed according to the treatment they actually received (ITT population). Median overall survival could not be estimated as most participants were living at the end of the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed/Cisplatin/Gefitinib | Pemetrexed/Cisplatin
Serious Adverse Events (participants affected / at risk) | 6/39 | 3/31
Other Adverse Events (participants affected / at risk) | 38/39 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin/Gefitinib (N=39) | Pemetrexed/Cisplatin (N=31)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Cisplatin/Gefitinib (N=39) | Pemetrexed/Cisplatin (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (12) | 3 (5)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (12) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 27 (63) | 20 (45)
Stomatitis (Gastrointestinal disorders) | 8 (13) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (52) | 15 (29)
Asthenia (General disorders) | 3 (5) | 1 (1)
Chest discomfort (General disorders) | 1 (2) | 2 (2)
Chest pain (General disorders) | 4 (4) | 3 (7)
Fatigue (General disorders) | 10 (20) | 5 (9)
Malaise (General disorders) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 2 (3) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 4 (5) | 0 (0)
Rhinitis (Infections and infestations) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (6) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 6 (7)
Creatinine renal clearance decreased (Investigations) | 3 (3) | 4 (8)
Haemoglobin decreased (Investigations) | 8 (8) | 11 (12)
Neutrophil count decreased (Investigations) | 8 (14) | 13 (26)
Weight decreased (Investigations) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 6 (9) | 8 (14)
Anorexia (Metabolism and nutrition disorders) | 19 (35) | 15 (24)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2)
Dizziness (Nervous system disorders) | 6 (8) | 3 (4)
Headache (Nervous system disorders) | 4 (6) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (8) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (12) | 4 (7)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (29) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 13 (21) | 6 (6)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Median overall survival cannot be estimated due to the high censor rate (25 participants per treatment group were censored). Most participants were still living at the end of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days